CLINICAL TRIAL: NCT00293345
Title: A Phase I Study of a Prolonged Infusion of Triapine in Combination With a Fixed Dose Rate of Gemcitabine in Patients With Advanced Solid Tumors and Lymphomas
Brief Title: 3-AP and Gemcitabine in Treating Patients With Advanced Solid Tumors or Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00119; NCI-2009-00119 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI-7043; OSU-2005C0031; CDR0000455043; OSU 05016 (Other: Ohio State University Medical Center); 7043 (Other: CTEP); U01CA076576 (NIH); NCT01645527 (obsolete NCT alias)
Record Dates: First submitted 2006-02-16; First posted 2006-02-17 (Estimated); Last update posted 2013-09-30 (Estimated); Status verified 2013-09

CONDITIONS: Anaplastic Large Cell Lymphoma; Angioimmunoblastic T-cell Lymphoma; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Intraocular Lymphoma; Nodal Marginal Zone B-cell Lymphoma; Primary Central Nervous System Hodgkin Lymphoma; Primary Central Nervous System Non-Hodgkin Lymphoma; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Hodgkin Lymphoma; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Adult T-cell Leukemia/Lymphoma; Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Mycosis Fungoides/Sezary Syndrome; Recurrent Small Lymphocytic Lymphoma; Small Intestine Lymphoma; Splenic Marginal Zone Lymphoma; Stage III Adult Burkitt Lymphoma; Stage III Adult Diffuse Large Cell Lymphoma; Stage III Adult Diffuse Mixed Cell Lymphoma; Stage III Adult Diffuse Small Cleaved Cell Lymphoma; Stage III Adult Hodgkin Lymphoma; Stage III Adult Immunoblastic Large Cell Lymphoma; Stage III Adult Lymphoblastic Lymphoma; Stage III Adult T-cell Leukemia/Lymphoma; Stage III Cutaneous T-cell Non-Hodgkin Lymphoma; Stage III Grade 1 Follicular Lymphoma; Stage III Grade 2 Follicular Lymphoma; Stage III Grade 3 Follicular Lymphoma; Stage III Mantle Cell Lymphoma; Stage III Marginal Zone Lymphoma; Stage III Mycosis Fungoides/Sezary Syndrome; Stage III Small Lymphocytic Lymphoma; Stage IV Adult Burkitt Lymphoma; Stage IV Adult Diffuse Large Cell Lymphoma; Stage IV Adult Diffuse Mixed Cell Lymphoma; Stage IV Adult Diffuse Small Cleaved Cell Lymphoma; Stage IV Adult Hodgkin Lymphoma; Stage IV Adult Immunoblastic Large Cell Lymphoma; Stage IV Adult Lymphoblastic Lymphoma; Stage IV Adult T-cell Leukemia/Lymphoma; Stage IV Cutaneous T-cell Non-Hodgkin Lymphoma; Stage IV Grade 1 Follicular Lymphoma; Stage IV Grade 2 Follicular Lymphoma; Stage IV Grade 3 Follicular Lymphoma; Stage IV Mantle Cell Lymphoma; Stage IV Marginal Zone Lymphoma; Stage IV Mycosis Fungoides/Sezary Syndrome; Stage IV Small Lymphocytic Lymphoma; Unspecified Adult Solid Tumor, Protocol Specific; Waldenström Macroglobulinemia
MeSH Terms: conditions — Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Intraocular Lymphoma; Lymphoma, B-Cell, Marginal Zone; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Leukemia, Lymphocytic, Chronic, B-Cell; Waldenstrom Macroglobulinemia | interventions — Gemcitabine; 3-aminopyridine-2-carboxaldehyde thiosemicarbazone

ARMS (1):
- Treatment (gemcitabine hydrochloride, triapine) (Experimental): Patients receive 3-AP (TriapineÃÂ®) IV over 24 hours followed by gemcitabine hydrochloride IV over 100-125 minutes on days 1 and 8. Treatment repeats every 3 weeks for 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: gemcitabine hydrochloride; Drug: triapine

INTERVENTIONS:
Drug: gemcitabine hydrochloride
  Other Names: dFdC; difluorodeoxycytidine hydrochloride; gemcitabine; Gemzar
Drug: triapine
  Other Names: 3-AP; OCX-191

SUMMARY:
This phase I trial is studying the best dose of 3-AP and the side effects of giving 3-AP together with gemcitabine in treating patients with advanced solid tumors or lymphoma. Drugs used in chemotherapy, such as 3-AP and gemcitabine (GEM), work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. 3-AP may help gemcitabine kill more cancer cells by making the cells more sensitive to the drug. 3-AP may also stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximal tolerable dose (MTD) of 3-AP administered as a 24 hour infusion in combination with and fixed-dose gemcitabine hydrochloride (GEM) in patients with advanced solid tumors or lymphomas.

SECONDARY OBJECTIVES:

I. To define the qualitative and quantitative toxicities of the 3-AP/GEM combination in regard to organ specificity, time course, predictability, and reversibility.

II. To document the therapeutic response of this combination in those patients when possible.

III. To measure deoxycytidine triphosphate (dCTP) levels in peripheral blood mononuclear cells (PBMCs) before and after treatment at specified times and try to correlate findings to activity and toxicity of 3-AP.

IV. To perform limited pharmacokinetic analysis.

OUTLINE: This is a dose-escalation study of 3-AP (Triapine®).Patients receive 3-AP (Triapine®) IV over 24 hours followed by gemcitabine hydrochloride IV over 100-125 minutes on days 1 and 8. Treatment repeats every 3 weeks for 12 courses in the absence of disease progression or unacceptable toxicity.

Patients achieving complete response (CR) receive 1 additional course of therapy beyond documented CR.Cohorts of 3-6 patients receive escalating doses of 3-AP (Triapine®) until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.After completion of study treatment, patients are followed periodically for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed advanced solid tumors or lymphoma

  * Disease considered incurable using standard treatment
* ECOG performance status ≤ 2
* Life expectancy > 12 weeks
* WBC ≥ 3,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Total bilirubin normal
* AST/ALT ≤ 2.5 times upper limit of normal
* Creatinine normal OR creatinine clearance ≥ 60 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception prior to and during study treatment
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to 3-AP (Triapine®) and/or gemcitabine hydrochloride
* No known glucose-6-phosphate dehydrogenase (G6PD) deficiency
* No uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situation that would limit compliance with study requirements
* No pulmonary disease (e.g., dyspnea at rest, supplemental oxygen requirement, or baseline oxygen saturation < 92%)
* Prior gemcitabine hydrochloride allowed if given as a standard 30-minute infusion

  * At least 4 weeks since prior gemcitabine hydrochloride
* Patient may have received < 2 lines of chemotherapy in the metastatic setting
* No prior 3-AP (Triapine®) or fixed-dose gemcitabine hydrochloride
* At least 6 weeks since prior nitrosoureas or mitomycin C
* More than 3 weeks since prior radiotherapy
* No other concurrent investigational agents
* No concurrent combination antiretroviral therapy in HIV-positive patients
* No other concurrent anticancer agents or therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-06; Primary Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
MTD as assessed by the number of patients with dose-limiting toxicity (DLT) | Observed clinically for 4 hours after each 3-AP infusion during the first cycle of treatment
  MTD is the maximum dose level with fewer than 2 of 3/6 patients experiencing DLT. The study uses standard method phase I design of dose escalation. DLT will be defined as greater or equal to Grade 3 non-hematologic or greater or equal to Grade 4 hematologic adverse event EXCEPT: greater or equal to Grade 3 nausea and greater or equal to Grade 3 vomiting that improves with antiemetic therapy; greater or equal to Grade 3 diarrhea that improves with Lomotil; and greater or equal to Grade 4 Neutropenia that recovers to less or equal to Grade 3 within 7 days of first identification.

SECONDARY OUTCOMES:
Toxicity as assessed using the NCI Common Toxicity Criteria, Version 3.0 | Observed clinically for 4 hours after each 3-AP infusion during the first cycle of treatment and monitored until disease progression or for a maximum of 24 months following termination of treatment
  Toxicities include neutropenia grade 4 (<500/mm3), neutropenic fever (grade 4 neutropenia and greater than or equal to grade 2 fever), thrombocytopenia Grade 3-4 (<50000/mm3), and non-hematologic toxicities grades 3-4. The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 will be utilized for adverse event reporting.
Therapeutic response | Tumor and radiologic measurements every 8 weeks from start of treatment. In addition to a baseline scan, confirmatory scans will also be obtained 8 weeks following initial documentation of an objective response.
  Response and progression will be evaluated in this study using the new international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) Committee. Complete Response (CR) is the disappearance of all target lesions. Partial Response (PR) requires at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD. The results will be purely descriptive.
Duration of overall response | Baseline until disease progression or for a maximum of 24 months following termination of treatment.
  The duration of overall response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started).
Duration of stable disease | Baseline until disease progression or for a maximum of 24 months following termination of treatment.
  Stable disease is measured from the start of the treatment until the criteria for progression are met, taking as reference the smallest measurements recorded since the treatment started.
Levels of dCTP in PBMCs correlated to activity and toxicity of 3-AP | PMBCs isolated immediately before and after 3-AP infusion (day 1), but before GEM is started on (day 2) on both course 1 and course 2 of treatment
  If dCTP levels are diminished by 3-AP, there is a real possibility of ribonucleotide reductase (RR) inhibition in tumor cells with a higher growth fraction (known to have elevated RR levels). It will also be possible to correlate the steady state levels of 3-AP with the concentration of dCTP in circulating cells. The RT-PCR of PBMCs before and after infusion would be helpful to reassure that the change of dCTP pool is correlated with 3-AP inhibiting RR.
Pharmacokinetics as assessed by steady state concentration (Css) of 3-AP in serum | On the first day of infusion (course 1 only) during the last 4 hours of 3-AP infusion

CONTACTS AND LOCATIONS:
Overall Officials: Tanios Bekaii-Saab, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States